CLINICAL TRIAL: NCT05607017
Title: The Role of Losartan in the Prevention of Early Structural Changes Associated With Radiation-Induced Heart Failure
Brief Title: Losartan in Prevention of Radiation-Induced Heart Failure
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rachel Beth Jimenez, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-457
Record Dates: First submitted 2022-11-01; First posted 2022-11-07 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Myocardial Fibrosis; Radiation-Induced Fibrosis
Keywords: Breast Cancer; Myocardial Fibrosis; Radiation-Induced Fibrosis
MeSH Terms: conditions — Breast Neoplasms; Radiation Fibrosis Syndrome | interventions — Losartan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Radiation Therapy and Losartan (Experimental): Participants will receive radiation therapy 5x weekly over 1-6 weeks. Participants will receive Losartan 1x daily during radiation therapy and for up to 6 months afterward then be followed for 1 year
  Interventions: Drug: Losartan; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Losartan — Taken Orally
  Other Names: Losartan Potassium
Radiation: Radiation Therapy — Photon Radiation Therapy

SUMMARY:
This study is being done to see if losartan affects the chances of developing radiation-induced heart failure in patients who are receiving radiation therapy as part of standard of care treatment for breast cancer.

The interventions involved in this study are:

* Losartan
* Radiation Therapy (standard of care)

DETAILED DESCRIPTION:
This is a pilot study examining whether losartan prevents radiation therapy-induced myocardial fibrosis (thickening of the heart tissue), which can cause heart failure, in breast cancer patients receiving radiation therapy.

Losartan is an U.S. Food and Drug Administration (FDA) approved drug used to treat hypertension (high blood pressure) and heart failure. The U.S. Food and Drug Administration (FDA) has not approved losartan for use in the treatment of breast cancer.

The FDA has approved radiation therapy as a treatment option for breast cancer.

The research study procedures include: screening for eligibility and study treatment including evaluations and follow up visits. It is expected participants will be on the study for 1 year.

It is expected that about 10 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

->18 years of age

* Non-metastatic Breast Cancer patients who are scheduled to receive conventional left breast/chest wall RT inclusive of treatment to the internal mammary lymph nodes (IMNs)
* Prior chemotherapy is permitted
* Patients must have Left-sided Breast Cancer
* Ability to understand and the willingness to sign a written informed consent document
* No contraindication to MRI

Exclusion Criteria:

* Person who is pregnant or breastfeeding.
* Patient unable to swallow oral medication.
* Patients receiving any other investigational agent will not be excluded from study eligibility, unless the patient is already enrolled in an interventional study evaluating cardiac toxicity
* Patients already receiving ACE/ARBs.
* Patients with a history of allergic reactions to Losartan biosimilars.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Extracellular Volume (ECV) of Myocardial Fibrosis | 6 months
  The primary endpoint is detectable decrease in extracellular volume as measured by cardiac MRI

SECONDARY OUTCOMES:
Serum cardiac biomarker | 6 months
  The secondary objective of this study is to compare pre- and post-Radiation Therapy changes in serum TGF-β levels

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jimenez, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation